CLINICAL TRIAL: NCT01864356
Title: A Randomized, Double Blind, Multi-Center, Placebo Controlled Study To Evaluate The Efficacy, Safety, And Tolerability Of Multiple Doses Of NT100 Following IVF In Women With A History Of Repeated IVF Failures (Thrive-IVF)
Brief Title: A Multi-Center Study To Evaluate Multiple Doses of NT100 Following IVF In Women With Repeated IVF Failures (Thrive-IVF)
Acronym: Thrive-IVF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nora Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NT-03
Record Dates: First submitted 2013-05-14; First posted 2013-05-29 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Repeated IVF Failure
Keywords: IVF failure; Repeated IVF failure; Implantation failure; Repeated implantation failure; IVF; NT100

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NT100 Dose 1 (Experimental): NT100 Dose 1
  Interventions: Drug: NT100
- NT100 Dose 2 (Experimental): NT100 Dose 2
  Interventions: Drug: NT100
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NT100
  Arms: NT100 Dose 1; NT100 Dose 2
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of multiple doses of subcutaneous NT100 vs placebo following in vitro fertilization (IVF) in women with a history of repeated IVF failures.

DETAILED DESCRIPTION:
NT-03 will be a randomized, double blind, multi-center, placebo controlled study of multiple doses of subcutaneous NT100 following IVF in women with a history of repeated IVF failures. Approximately 150 subjects will be randomized in a 1:1:1 ratio to receive subcutaneous NT100 low dose, NT100 high dose, or placebo, qd for up to 4 weeks.

Screening will include a standard IVF stimulation protocol, followed by fertilization and culture of embryos. If the subject remains eligible, she will be randomized to receive study drug. All subjects will be followed for 4 weeks after the last dose of study drug. At Week 10 of gestation, subjects who are pregnant will roll over into a follow-up study (NT-04) to assess subsequent pregnancy, delivery, and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female 21-38 years of age at screening
* History of repeated IVF failures despite transfer of good-quality embryos, defined as follows:
* ...1) 3 or more IVF cycles involving transfer of at least two good-quality cleavage-stage embryos or at least one good-quality blastocyst (2010 SART (Society for Assisted Reproductive Technologies) grading criteria)that resulted in one of the following outcomes:
* * .....a) no pregnancy
* * .....b) biochemical pregnancy
* * .....c) spontaneous abortion of an intrauterine clinical pregnancy before or equal to completed Week 8 of gestation
* ...2) At least two of the eligible IVF failures must have involved transfer of fresh embryos
* ...3) At least two of the eligible IVF failures must have involved retrieval of at least 5 oocytes
* ...4) No live birth, abortion later than Week 8 of gestation, or stillbirth may have occurred since the first of these IVF failures
* Body mass index (BMI) of 19-38 kg per m2 at screening
* TSH (thyroid-stimulating hormone) less than or equal to 4.0 mIU/L(milli-International units per Liter) for subjects with no history of hypothyroidism, or TSH less than or equal to 2.5 mIU/L for subjects with a history of hypothyroidism, at screening

Exclusion Criteria:

* Prior diagnosis of moderate or severe ovarian hyperstimulation syndrome (OHSS)
* Clinically confirmed polycystic ovary syndrome (PCOS)
* History of a major congenital anomaly in the subject, her current male partner, or first degree relative of either the subject or her current male partner
* Known karyotype abnormalities in either the subject or her current male partner / sperm donor
* Any prior pregnancy terminated for a fetal medical condition
* History of severe (stage IV) endometriosis
* Current or past systemic autoimmune disease
* Any uncontrolled clinically significant medical condition (e.g. asthma, Type II diabetes, infection)

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Ongoing clinical pregnancy rate | Week 8 of gestation
  The primary efficacy outcome measure is the ongoing clinical pregnancy rate at Week 8 of gestation.

SECONDARY OUTCOMES:
Biochemical evidence of pregnancy rate (as measured by hCG) | Week 4 of gestation
Ongoing clinical pregnancy rate | Weeks 6 and 10 of gestation
Implantation rate following embryo transfer | Week 8 of gestation
Number of subjects with adverse events and serious adverse events | through 4 weeks after last dose of study drug (up to Week 10 of gestation)
Changes in clinical laboratory parameters following study drug exposure | through 4 weeks after the last dose of study drug (up to Week 10 of gestation)
Moderate to severe ovarian hyperstimulation syndrome (OHSS) rate | through Week 10 of gestation

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - HRC Fertility, Encino, California
  - HRC Fertility, Newport Beach, California
  - HRC Fertility, Pasadena, California
  - UCSF, San Francisco, California
  - Reproductive Associates of Delaware, Newark, Delaware
  - Columbia Fertility Associates, Washington D.C., District of Columbia
  - Florida Fertility Institute, Clearwater, Florida
  - IVF and Fertility Center of Miami, Miami, Florida
  - Georgia Reproductive Specialists, Atlanta, Georgia
  - Fertility Centers of Illinois / River North IVF Center, Chicago, Illinois
  - Fertility Centers of Illinois / Highland Park IVF Center, Highland Park, Illinois
  - Shady Grove Fertility, Rockville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston IVF, Waltham, Massachusetts
  - Columbia University, New York, New York
  - Institute for Reproductive Health, Cincinnati, Ohio
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Center for Assisted Reproduction, Bedford, Texas
  - Houston Fertility Institute, Houston, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Utah Fertility Center, Pleasant Grove, Utah